CLINICAL TRIAL: NCT03362450
Title: Prenatal Diagnosis of Antenatal Midgut Volvulus: Specific Ultrasound Features
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0321
Record Dates: First submitted 2017-10-25; First posted 2017-12-05 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-10

CONDITIONS: Fetal Volvulus; Midgut Volvulus
Keywords: Midgut volvulus; Fetal volvulus; Whirlpool sign; Pregnant women; Position of mesenteric vessels; Post natal surgery; Foetopathology if performed; Hydro-meconium level in the dilated loops
MeSH Terms: conditions — Volvulus Of Midgut | interventions — Pregnancy Trimester, Third; Autopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant patients seen for second or third trimester: Foetus with diagnosis of prenatal volvulus based on post-natal findings and prenatal imaging findings
  Interventions: Other: Fetal ultrasound during the second or third trimester/ Postnatal surgery / Post mortem examination

INTERVENTIONS:
Other: Fetal ultrasound during the second or third trimester/ Postnatal surgery / Post mortem examination — Fetal ultrasound during the second or third trimester Postnatal surgery Post mortem examination

SUMMARY:
Objective:

The small bowel volvulus is a rare cause of intestinal obstruction which may occur in utero and whose prenatal diagnosis is difficult.Sonographic signs are mainly indirect and non specific.The aim of this study is to present a retrospective analysis of prenatal sonographicfindings in fetal segmental midgut volvulus.Thanks to this series the investigators could highlight the more specifics signs of the volvulus included a new pattern.

DETAILED DESCRIPTION:
Objective:

The small bowel volvulus is a rare cause of intestinal obstruction which may occur in utero and whose prenatal diagnosis is difficult. Sonographic signs are mainly indirect and nonspecific. The aim of this study is to present a retrospective analysis of prenatal sonographic findings in fetal segmental midgut volvulus. Thanks to this series the investigators could highlight the more specifics signs of the volvulus included a new pattern.

Methods:

Unicentric retrospective analysis of cases of prenatal midgut volvulus between 2006 and 2017. The primary inclusion criteria was postnatal diagnosis of prenatal volvulus based on post-natal findings and prenatal imaging findings. The exclusion criteria was the absence of prenatal imaging assessment. The investigators collected the clinical history and the echographic mode B and color Doppler. They have searched for some specific sign like " whirlpool sign " representing the winding of the mesenteric vein around the superior mesenteric arterywith color Doppler with arciform pattern of the midgut, hydro-meconium level in the dilated loops and position of mesenteric vessels for evaluation of the intestinal (mal) rotation. Gold standard was surgery or foetopathology if performed.

ELIGIBILITY:
Inclusion Criteria:

* postnatal diagnosis of prenatal volvulus based on post-natal findings and prenatal imaging findings

Exclusion Criteria:

* the absence of prenatal imaging assessment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — All pregnant women
Study Population: All pregnant women
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
echography | during the second (22-24 weeks) after ultrasound screening
  Observation of specific signs using echography for the diagnosis of fetal during the second (22-24 weeks) and the third (31-34 weeks) trimester after ultrasound screening and when diagnostic ultrasound were performedmidgut volvulus
echography | the third (31-34 weeks) trimester after ultrasound screening
  Observation of specific signs using echography for the diagnosis of fetal

SECONDARY OUTCOMES:
ultrasound signs of complication | the third (31-34 weeks) after ultrasound screening
  Observation of ultrasound signs of complication of midgut volvulus during the pregnancy like meconial pseudocyst, ascites, meconial peritonitis.
ultrasound signs of complication | during the second (22-24 weeks) after ultrasound screening
  Observation of ultrasound signs of complication of midgut volvulus during the pregnancy like meconial pseudocyst, ascites, meconial peritonitis.
ultrasound signs of complication | 1 day
  Observation of ultrasound signs of complication of midgut volvulus during the pregnancy like meconial pseudocyst, ascites, meconial peritonitis after diagnostic ultrasound.
ultrasound signs of complication | just after delivery
  Observation of ultrasound signs of complication of midgut volvulus during the pregnancy like meconial pseudocyst, ascites, meconial peritonitis.
presence or not of the volvulus | 1 day
  Observation of surgery outcome like presence or not of the volvulus after diagnostic ultrasound
presence or not of the volvulus | during the second (22-24 weeks) after ultrasound screening
  Observation of surgery outcome like presence or not of the volvulus
presence or not of the volvulus | just after delivery
  Observation of surgery outcome like presence or not of the volvulus
presence or not of the volvulus | the third (31-34 weeks) after ultrasound screening
  Observation of surgery outcome like presence or not of the volvulus
presence or not ileal atresia. | during the second (22-24 weeks) after ultrasound screening
  Observation of surgery outcome like presence or not ileal atresia
presence or not ileal atresia. | the third (31-34 weeks) after ultrasound screening
  Observation of surgery outcome like presence or not ileal atresia
presence or not ileal atresia. | just after delivery
  Observation of surgery outcome like presence or not ileal atresia
presence or not ileal atresia. | 1 day
  Observation of surgery outcome like presence or not ileal atresia after diagnostic ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Uhmontpellier, Montpellier, France